CLINICAL TRIAL: NCT06065722
Title: Akynzeo or Olanzapine for Patients Who Experience Breakthrough CINV in Patient Receiving Moderately or Highly Emetogenic Chemotherapy After First Cycle of Chemotherapy
Brief Title: Prevention of Breakthrough CINV in Patients Receiving Moderately or Highly Emetogenic Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simon Williamson Clinic (Industry)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SWC999
Record Dates: First submitted 2023-09-24; First posted 2023-10-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: chemotherapy induced nausea and vomiting; NK-1; olanzapine
MeSH Terms: conditions — Vomiting | interventions — netupitant, palosentron drug combination; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AKYNZEO for patient receiving MEC (Active Comparator): Add Akynzeo to 5HT3 And dexamethasone
  Interventions: Drug: Akynzeo
- oLANZAPINE and Akynzeo to patients receiving highly emetogenic (Active Comparator): olANZAPINE plus Akynzeo
  Interventions: Drug: Akynzeo

INTERVENTIONS:
Drug: Akynzeo — OLANZAPINE
  Other Names: Olanzapine

SUMMARY:
The purpose of the proposed study is to provide a clinical approach to chemotherapy induced nausea and vomiting (CINV) prophylaxis in cycle 2 of moderately emetogenic chemotherapy or highly emetogenic chemotherapy for patients who developed breakthrough CINV after cycle 1 based on the available data in the literature as well as the recommendations provided by established guidelines

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting (CINV) adversely affects patients' quality of life and may affect patients' treatment decisions. The emetogenicity of the chemotherapy administered and specific patient characteristics such as female gender, age, and history of low alcohol intake can increase a patients' risk for CINV.

Table 1. Patient-Related Risk Factors for Emesis Following Chemotherapy Major Factors Minor Factors Female History of Motion Sickness Age < 50 years Emesis during past pregnancy History of prior low chronic alcohol intake (<1 ounce of alcohol/day) Anxiety History of previous chemotherapy-induced emesis

Significant and uncontrolled CINV may result in patients returning to the chemotherapy treatment facility one to three days post-chemotherapy for rehydration, or emesis or nausea control. If CINV cannot be controlled in an outpatient facility, patients may subsequently be treated in an emergency department or require hospitalization. Patients who have an electrolyte imbalance or those who have recently undergone surgery or radiation therapy, are at greater risk of experiencing serious complications from CINV.

The use of 5-hydroxytryptamine-3 (5-HT3) receptor antagonists has improved the control of CINV Additional improvement in the control of CINV has occurred with the use of neurokinin-1 (NK-1) receptor antagonists, and olanzapine, an antipsychotic which blocks multiple neurotransmitters in the central nervous system.

The primary endpoint used for studies evaluating various agents for the control of CINV has been complete response (CR) (no emesis, no use of rescue medication) over the acute (24 hours post-chemotherapy), delayed (24-120 hours), and overall (0-120 hours) periods. The combination of a 5-HT3 receptor antagonist, dexamethasone, and a NK-1 receptor antagonist have improved the control of emesis in patients receiving either highly emetogenic chemotherapy (HEC) or moderately emetogenic chemotherapy (MEC) over a 120-hour period following chemotherapy administration

The use of effective antiemetic agents in various clinical settings has been described in established guidelines from the Multinational Association of Supportive Care in Cancer (MASCC) and the European Society of Medical Oncology (ESMO), the American Society of Clinical Oncology (ASCO)], and the National Comprehensive Cancer Network (NCCN).

The purpose of the proposed is to provide a clinical approach to CINV prophylaxis in cycle 2 of MEC or HEC for patients who developed breakthrough CINV after cycle 1 based on the available data in the literature as well as the recommendations provided by established guidelines.

ELIGIBILITY:
Inclusion Criteria:

* CHEMOTHERAPY NAIIVE
* patient receiving moderately or highly emetogenic chemotherapy
* lung cancer
* breast cancer

Exclusion Criteria:

* PRIOR CHEMOTHERAPY for any cancer
* nausea or vomiting 24 hours prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
COMPELETE RESPONSE, no vomiting or use of rescue medications | 5 DAYS post chemotherapy
  No vomiting or use of rescue medications for 5 days post chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Rudolph M Navari, Mount Olive, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navari RM, Bonizzoni E. NEPA (Netupitant/Palonosetron) for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Patients Receiving Highly or Moderately Emetogenic Chemotherapy Who Experienced Breakthrough CINV in Cycle 1 of Chemotherapy: A Phase II Clinical Trial. Cancer Med. 2025 Apr;14(7):e70549. doi: 10.1002/cam4.70549. PMID 40145359